CLINICAL TRIAL: NCT06578845
Title: HappyMums - Can Data Collected by a Mobile App be Used to Help Learn More About Mental Health Symptoms in Pregnant Women and Birthing People at Risk of Depression in Pregnancy?
Brief Title: HappyMums Mobile Application Study
Acronym: HappyMums
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: University of Milan (Other); Ospedale San Raffaele (Other); Catholic University of Croatia (Unknown); University of Helsinki (Other); Charite University, Berlin, Germany (Other); SWPS University of Social Sciences and Humanities (Other); Ab.Acus (Other); University of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: KCL IRAS 339391
Record Dates: First submitted 2024-05-28; First posted 2024-08-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Antenatal Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant people currently experiencing, or at risk of, antenatal depression: All eligible participants will be given access to the 'HappyMums' mobile application, which will be used to collect data pertinent to their mental health status during pregnancy.

SUMMARY:
The goal of this study is to investigate whether pregnant people at risk of, or currently suffering from antenatal depression, find it acceptable to use the 'HappyMums' mobile application during their pregnancy. This app will collect data relevant to their mental health passively and through active engagement from the user. After the study is complete, these data will be put together to determine if such data types could be used in future to help predict and identify antenatal depression, and aid better treatment decisions.

DETAILED DESCRIPTION:
HappyMums aims to develop a digital platform (smartphone app), and investigate whether data collected by a mobile app can be used to help learn more about mental health symptoms in pregnant women and birthing people at risk of depression in pregnancy.

This study aims to investigate the acceptability and usability of the HappyMums App. Following data collection, data will be aggregated to generate statistical models, with the aim of testing their predictive ability for antenatal depression trajectories.

The application will collect and integrate heterogenous data and will also allow an improvement of lifestyle attitudes, the maintenance of wellbeing in pregnancy, and the continuous monitoring of treatment efficacy. HM will therefore contribute to reducing the stigma by empowering mothers and birthing parents to monitor and master their mental health.

The study objective is to actively and passively gather data relevant to perinatal mental health, via a mobile application, which will be used to retrospectively develop an algorithm capable of identifying mental health trajectories in at-risk women/birthing people. The app will include game-like activities, access to an antenatal wellbeing course and space for pregnancy- and health-related data logging and monitoring. It will also utilise smartphone sensors to collect passive data types such as GPS, phone usage and step counts. This study will test the use of such mobile applications for patient mental health monitoring, and will also collect traditional research data such as biological samples and standardised questionnaires to be used as comparators to app-derived data.

Participants: Participants will be pregnant people either currently experiencing depressive symptoms, or who meet criteria for at least one risk factor for antenatal depression, previously identified from the literature, such as pregnancy complications or lack of social support. They will be recruited from 13 weeks' gestation to 28 weeks' gestation.

Recruitment: Recruitment will be conducted through self-referral, social media and online advertisement, and poster/flyer advertising in spaces and publications relevant to pregnant people, such as antenatal and health clinics, antenatal education spaces, children and family centres and newsletters.

Measures and Outcomes: Models will be generated to determine the ability of passively and actively app-collected data to predict antenatal depression symptoms through pregnancy, and how this compares to traditional measures such as standardised mental health questionnaires: Edinburgh Postnatal Depression Scale (EPDS), Generalised Anxiety Disorder Assessment (GAD-7) and Patient Health Questionnaire (PHQ-9).

For further cohort characterisation and to determine the influence of risk factors, other measures will also be collected and tested in the model: Mini International Neuropsychiatric Interview (subset only), Childhood Trauma Questionnaire (subset only), Adult Attachment Questionnaire, Life Events, Composite Abuse Scale, Maternal Antenatal Attachment Scale (subset only), Perceived Stress Scale (subset only), Multidimensional Scale of Perceived Social Support (subset only), Couple Satisfaction Index (subset only) and Postpartum Bonding Questionnaire (subset only).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people, aged 18 or older and up to 28 weeks' gestation.
* Satisfactory understanding of English/national language of host country, in order to give fully informed consent.
* Either suffering with depressive symptoms currently, or who have at least one risk factor for antenatal depression.
* Owning a smartphone capable of downloading and running HappyMums application

Exclusion Criteria:

* Inability to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will consist of pregnant participants, up to 28 weeks' gestation, who have at least one risk factor for antenatal depression, or current depressive symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who continue to use mobile application from enrolment until they give birth. | From enrolment to end of pregnancy.
  The primary outcome is whether participants feel able to continue to use the app throughout their pregnancy. Usage data of the app will be logged to ascertain if participants continue to engage with it throughout their pregnancy. 'Usage' of the application will be defined as submission of any questionnaire, logging of data, or interaction with any other activities or content on the application. This will be quantified as proportion of participants who use the app weekly from their enrolment on the app to the end of their pregnancy.

SECONDARY OUTCOMES:
Usability of the mobile application - System Usability Scale | Administered once - to be completed from delivery to 2 months postpartum.
  Questionnaire given to participants after pregnancy to ascertain if they find the app system usable.
Acceptance of the mobile application - Unified Theory of Acceptance and Use of Technology Scale. | Administered once - to be completed from delivery to 2 months postpartum.
  Questionnaire given to participants after pregnancy to ascertain if they find the app system acceptable.
Severity of antenatal depression - Edinburgh Postnatal Depression Scale | Every 2 weeks from enrolment to end of pregnancy.
  Antenatal depression will be measured using the EPDS, and will be available to complete on the application every 2 weeks.
Development of clinically significant depression - Mini International Neuropsychiatric Interview | Administered at enrolment and up to 2 months postpartum
  The MINI will be administered to a validation sub-cohort to identify development of, or change in, symptoms of Major Depressive Disorder. This will be used to validate app-derived data types used to identify depression.

CONTACTS AND LOCATIONS:
Locations (7):
- Catholic University of Croatia, Zagreb, Croatia
- University of Helsinki, Helsinki, Finland
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Italy (2):
  - San Raffaele Hospital, Milan
  - University of Milan, Milan
- SWPS University, Warsaw, Poland
- King's College London, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Priestley K, Laijawala R, Hazelgrove K, Bind R, Rebecchini L, Mariani N, Alford S, Kirkpatrick M, Mancino F, Kim S, Pushpakanthan S, Biaggi A, Cavaliere L, Di Benedetto MG, Matijas M, Zutic M, Brekalo M, Nakic Rados S, Zukowska K, Braniecka A, Jackowska M, Bessi M, Agnoletto E, Melloni EMT, Benedetti F, Bulgheroni M, La Gamba M, Martin Isla C, Izquierdo Morcillo C, Lekadir K, Salo V, Seikku T, Raikkonen K, Godara M, Schneider-Schmid UM, Entringer S, Buss C, de Barra D, Woods A, Dazzan P, Cattaneo A, Pariante C. HappyMums mobile application study protocol: use of a smartphone application to gather data predictive of antenatal depression. BMJ Open. 2026 Feb 4;16(2):e106978. doi: 10.1136/bmjopen-2025-106978. PMID 41638734